CLINICAL TRIAL: NCT05691647
Title: Chronotherapy for Patients With a Depressive Episode in a Public Mental Health Care Clinic in Norway: A Randomized Controlled Trial
Brief Title: Chronotherapy for Depressive Episodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 480812
Record Dates: First submitted 2022-12-16; First posted 2023-01-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Depressive Episode
MeSH Terms: interventions — Chronotherapy; Therapeutics

STUDY DESIGN:
Masking Description: Masking will not be applicable due to the nature of the study, in which participants randomized to receive chronotherapy plus treatment as usual will be admitted to the ward for a one-night sleep deprivation, and the participants and researchers will understand which intervention arm the participant is receiving. Researchers and participants will not be aware of randomization until after baseline-assessments are completed. Analyses will be conducted by a statistician who is blinded to intervention allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronotherapy + treatment as usual (Experimental)
  Interventions: Behavioral: Chronotherapy; Behavioral: Treatment as usual
- Treatment as usual (Active Comparator): medication, cognitive behavioral therapy, and other psychotherapies.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Chronotherapy — Chronotherapy involves three different interventions. Sleep deprivation/wake therapy will be conducted for 34 hours. To assist wake and to ensure that the participants adhere to the sleep deprivation, outpatients will be admitted to a one-night stay at the inpatient ward that is connected to the outpatient clinic at Nidaros DPS. Patients already admitted to inpatient treatment will be temporary transferred to the ward selected to oversee the sleep deprivation. Upon discharge, participants are encouraged to adhere to the sleep schedule which presents the sleep-wake phase advancement and later stabilization of the sleep-wake phase. Light therapy is provided for half an hour every day from day four in the study. In addition to the chronotherapeutic interventions, the participants will receive treatment as usual (TAU) with their assigned therapist.
  Arms: Chronotherapy + treatment as usual
Behavioral: Treatment as usual — Participants allocated to receive TAU alone, will receive standard treatment for a depressive episode in the outpatient or the inpatient clinic. This study will not give restrictions or guidelines on how this treatment should be performed. The TAU-group will receive the treatment the responsible therapist considers and evaluate best fitting in the situation. Typical interventions administered in therapy for a depressive episode includes medication, cognitive behavioral therapy, and other psychotherapies.

SUMMARY:
Evidence-based treatments for depression, such as antidepressive medication, usually have a latency of 4 to 6 weeks before they achieve a therapeutic effect. Chronotherapy is a group of non-pharmacological interventions that presumably act on the circadian system to achieve a rapid-onset clinical effect and better long-term effects and has been shown efficient to improve depressive symptoms. Interventions include sleep deprivation, sleep-phase advancement and stabilization, and light therapy. There are few studies testing the effectiveness of combining these three chronotherapeutic techniques in the initial phase of treatment of depression in a mental health care clinic. The investigators aim to test the effects and safety of chronotherapy in addition to TAU compared to TAU alone, with the primary outcome being self-reported depressive symptoms at 1 week following randomization. The study is a randomized controlled trial with 76 patients with a depressive episode who initiate treatment at Nidaros DPS, St. Olavs University Hospital. Participants will be allocated 1:1 to either chronotherapy + treatment as usual (TAU) or to TAU alone.

ELIGIBILITY:
Inclusion criteria. Patients eligible for the trial must comply with all the following at randomization:

* Being 18 years or older
* Willing and able to provide a written informed consent
* Newly diagnosed with an ongoing moderate or severe depressive episode according to the International Classification of Disorders 10th edition (ICD-10) and accepted for treatment for the depressive episode. The diagnosis is set in consensus of a licensed therapist and a specialist in psychiatry/psychology.
* The patient must score ≥ 9 on the Hamilton Depression Rating Scale-6.
* Must be able to communicate in a Scandinavian language

Exclusion criteria. Patients are considered ineligible for participation if any of the following are present:

* Illnesses and treatments where chronotherapy may be contraindicated (for example epilepsy, ongoing attack of multiple sclerosis, blindness, narcolepsy and psychotic depression, ECT treatment).
* Known pregnancy.
* Individuals with a known diagnosis of emotionally unstable personality disorder (F60.3).
* Individuals with a known psychotic disorder
* Shiftwork or other related social or work circumstances that inhibit participation
* Participation in an ongoing trial at the outpatient clinic that encompasses digital cognitive behavior therapy for insomnia (recruitment to this trial will end in 2023).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in self-reported levels of depressive symptoms at week 1 after randomization | 1 week after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.

SECONDARY OUTCOMES:
Between-group difference in observer-rated levels of depressive symptoms at week 1 after randomization. | 1 week after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in observer-rated levels of depressive symptoms at week 2 after randomization | 2 weeks after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in observer-rated levels of depressive symptoms at week 4 after randomization. | 4 weeks after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in observer-rated levels of depressive symptoms at week 8 after randomization | 8 weeks after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in observer-rated levels of depressive symptoms at week 24 after randomization | 24 weeks after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in observer-rated levels of depressive symptoms at week 52 after randomization | 52 weeks after randomization
  Assessed with the Hamilton Depression Rating Scale (HDRS-6), a 6-item questionnaire for depressive symptoms the last 24 hours. Each item is rated on a 0 to 4 rating scale with higher scores indicating more depressive symptoms. The range is 0-22.
Between-group difference in self-reported anxiety symptoms at week 1 after randomization | 1 week after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported anxiety symptoms at week 2 after randomization. | 2 weeks after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported anxiety symptoms at week 4 after randomization | 4 weeks after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported anxiety symptoms at week 8 after randomization | 8 weeks after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported anxiety symptoms at week 24 after randomization | 24 weeks after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported anxiety symptoms at week 52 after randomization | 52 weeks after randomization
  Here assessed with the General Anxiety Disorder (GAD-7), a 7 items self-report scale for central symptoms of anxiety over the last 14 days. The range is 0 to 21, with higher scores indicating more severe anxiety.
Between-group difference in self-reported insomnia symptoms at week 1 after randomization | 1 week after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in self-reported insomnia symptoms at week 2 after randomization. | 2 weeks after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in self-reported insomnia symptoms at week 4 after randomization | 4 weeks after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in self-reported insomnia symptoms at week 8 after randomization | 8 weeks after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in self-reported insomnia symptoms at week 24 after randomization | 24 weeks after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Between-group difference in self-reported insomnia symptoms at week 52 after randomization. | 52 weeks after randomization
  Here assessed with the Insomnia Severity Index (ISI), a 7-item questionnaire for the severity of insomnia symptoms the last 14 days. Each item is rated on a 0 to 4 rating scale with higher scores indicating more severe symptoms. The ISI has good psychometric properties and is validated for online use. Range is 0-28 with higher values represent higher levels of insomnia symptom severity.
Prospective daily sleep-wake pattern at day 3 after randomization | 3 days after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at day 4 after randomization. | 4 days after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 1 after randomization. | 1 week after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 2 after randomization. | 2 weeks after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 4 after randomization. | 4 weeks after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 8 after randomization | 8 weeks after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 24 after randomization. | 24 weeks after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Prospective daily sleep-wake pattern at week 52 after randomization | 52 weeks after randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.
Chronotype at week 8 after randomization. | 8 weeks after randomization
  Here assessed with the Reduced Morningness - Eveningness Questionnaire (rMEQ), a widely used measure of chronotype i.e. time preference for daily activities, including bed-times. The rMEQ has five items yielding scores from 4 to 25, with lower scores indicating "eveningness" and higher scores indicating "morningness". Higher scores indicate higher levels of morningness. Scores can be divided into five categories: definitely evening type (score <8), moderately evening type (Score 8-11), neither type (score 12-17), moderately evening type (score 18-21), and definitely morning type (score >21).
Work and social adjustment at week 1. | 1 week after randomization.
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
Work and social adjustment at week 2. | 2 weeks after randomization.
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
Work and social adjustment at week 4. | 4 weeks after randomization
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
Work and social adjustment at week 8. | 8 weeks after randomization
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
Work and social adjustment at week 24 | 24 weeks after randomization
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
Work and social adjustment at week 52 | 52 weeks after randomization
  Assessed with the Work and Social Adjustment Scale (WSAS). WSAS is a self-administered questionnaire that measures the subjective experience of functionality in work and social environments. The 5 items are rated on an 8-point Likert scale. Total scores range from 0-40, with a higher score indicating more functional impairment.
General health and health-related quality of life at week 1 | 1 week after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
General health and health-related quality of life at week 2. | 2 weeks after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
General health and health-related quality of life at week 4. | 4 weeks after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
General health and health-related quality of life at week 8 | 8 weeks after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
General health and health-related quality of life at week 24 | 24 weeks after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
General health and health-related quality of life at week 52. | 52 weeks after randomization.
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Patient satisfaction and experienced negative effects at week 4 after randomization | 4 weeks after randomization.
  A self-report measure was developed to assess the subjective experiences of patients in the study. The measure includes items to assess whether there have been positive and negative effects of the interventions and will include a free-text space to elaborate if none of the expected effects are experienced.
Serious adverse events will be assessed after 52 weeks after randomization. | 52 weeks after randomization.
  Adverse events will be reported to the study team continuously throughout the study period, and will be registered. Any serious adverse events will be reported.
Use of health care services at 52 weeks after randomization. | 52 weeks after randomization
  Assessed through questionnaires and health care records.
Use of health care services at 5 years after randomization | 5 years after randomization
  Assessed through questionnaires and health care records.
Use of health care services at 10 years after randomization. | 10 years after randomization.
  Assessed through questionnaires and health care records.
Between-group difference in self-reported levels of depressive symptoms at day 3 after randomization | 3 days after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Between-group difference in self-reported levels of depressive symptoms at day 4 after randomization | 4 days after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84. On day 4, sleep items will be excluded from the questionnaire.
Between-group difference in self-reported levels of depressive symptoms at week 2 after randomization | 14 days after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Between-group difference in self-reported levels of depressive symptoms at week 4 after randomization | 4 weeks after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Between-group difference in self-reported levels of depressive symptoms at week 8 after randomization | 8 weeks after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Between-group difference in self-reported levels of depressive symptoms at week 24 after randomization | 24 weeks after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Between-group difference in self-reported levels of depressive symptoms at week 52 after randomization | 52 weeks after randomization
  Assessed with the Inventory of Depressive Symptomatology Self-Report (IDS-SR), a 30-item questionnaire assessing depressive symptomatology. Items are rated on a Likert scale from 0 to 3, with higher scores indicating more depressive symptoms. The range is 0-84.
Subjective sleepiness during sleep deprivation | Day 3-4 after randomization
  Assessed with the Karolinska Sleepiness Scale (KSS), a 9-item Likert scale, scored from 1 (=extremely alert) to 9 (=extremely sleepy-fighting sleep). The assessment will take place every second hour during the sleep deprivation for the intervention group.
Expectations to the interventions at baseline | Day 0 after randomization
  Assessed with the Stanford Expectations of Treatment Scale (SETS), a 6-item questionnaire that assesses participants' positive and negative expectations to the interventions on a Likert scale from 1 (strongly disagree) to 7 (strongly agree)
Quality-adjusted life years (QALY) at week 1 after randomization | Week 1 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Quality-adjusted life years (QALY) at week 2 after randomization | Week 2 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Quality-adjusted life years (QALY) at week 4 after randomization | Week 4 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Quality-adjusted life years (QALY) at week 8 after randomization | Week 8 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Quality-adjusted life years (QALY) at week 24 after randomization | Week 24 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Quality-adjusted life years (QALY) at week 52 after randomization | Week 52 after randomization
  Assessed with the EQ-5D-5L. The EQ-5D-5L is a self-administered questionnaire that assesses general health and health-related quality of life at the day of measurement. The 5 items are rated on a 5-point Likert scale in addition to a 0-100 rating of overall experienced health condition.
Prospective daily sleep-wake pattern at day -7 before randomization. | Day -7 before randomization.
  Here assessed with the Consensus Sleep Dairy and actigraphy, which will be completed by the participant at baseline and each follow-up point for 14 days.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olavs Hospital, Nidaros DPS, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that underlie the results will be available after publication of the final version of the trial to researchers from accredited research institutions. Access to data will be limited to investigators who provide a methodologically sound proposal and will be for a specified time period (commencing about 3 months after publication and ending after five years). To ensure GDPR compliance, data processing must be covered by the 'Standard Contractual Clauses' from the European Commission, that data requesters have to sign. Proposals and requests for data access should be directed to the principal investigator.

REFERENCES:
- [Derived] Ramfjord LS, Kahn N, Langsrud K, Halvorsen JOO, Morken G, Saksvik S, Engvik LSS, Lydersen S, Kallestad H. Chronotherapy for patients with a depressive episode treated in a public outpatient mental healthcare clinic in Norway: protocol for a randomised controlled trial. BMJ Open. 2024 Jan 3;14(1):e076039. doi: 10.1136/bmjopen-2023-076039. PMID 38171633